CLINICAL TRIAL: NCT03666377
Title: The Impact of Chewing Gum on Postoperative Ileus in Children Who Undergo Abdominal Surgery: a Prospective, Randomized, Controlled Pilot Study
Brief Title: Chewing Gum on Postoperative Ileus in Children
Acronym: GUM_1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Anna Shawyer, Pediatric Surgeon, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2018:008
Record Dates: First submitted 2018-03-16; First posted 2018-09-11 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Bowel Ileus; Flatus
MeSH Terms: conditions — Ileus; Flatulence | interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomized, controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No gum chewing (No Intervention): Usual pharmacologic treatment and post-operative care (e.g. daily visits by surgical team, antibiotics where appropriate, mobilization, advancement of diet as tolerated). Analgesia and anti-emetics will be provided (both oral and intravenous) as needed.
- Gum chewing (Experimental): Usual pharmacologic treatment and post-operative care (e.g. daily visits by surgical team, antibiotics where appropriate, mobilization, advancement of diet as tolerated). Analgesia and anti-emetics will be provided (both oral and intravenous) as needed.
  Intervention: 1 piece of sugarless gum to be chewed three times daily for 1 hour each.
  Interventions: Other: Gum chewing

INTERVENTIONS:
Other: Gum chewing — 1 piece of sugarless gum to be chewed three times daily for 1 hour each.
  Arms: Gum chewing

SUMMARY:
Traditional postoperative care has been challenged recently to improve and speedup recovery (including the return of bowel function) such that patients can be discharged to home more quickly. This approach includes earlier mobilization of the patient, and introducing solid food sooner. Additionally, there is evidence in adults to suggest that "sham feeding" by chewing gum may also speed up bowel recovery so the patient may tolerate a solid diet earlier.

The aim of this study is to determine if gum chewing can enhance bowel recovery in children who undergo abdominal surgery.

DETAILED DESCRIPTION:
After intestinal surgery, many patients suffer from a "postoperative ileus" (POI). The cause is multifactorial and can be attributed to surgery itself, the lingering effect of the anesthetic, the use of narcotics and decreased mobility of the patient.

An ileus can delay the time to full diet, thus lengthening the hospital stay of the patient - sometimes up to several weeks.

There is evidence that early drinking/eating and increased mobility may accelerate the return of bowel function. "Fast-tracking" is well documented in the adult literature; protocols have been put in place to enhance GI tract recovery and thus decrease the morbidity of a prolonged hospital stay and ileus. "Fast-tracking" has been done in pediatric patients but not in a large RCT for abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children more than or equal to 4 years of age
* Children who undergo abdominal surgery (both laparoscopic or open)
* Children who have an expected postoperative length of stay more than 24 hours

Exclusion Criteria:

* Children who are less than 4 years of age
* Children who are unable to chew gum/swallow (e.g. intubated, decreased level of consciousness, cognitive or physical disability)
* Children or their parents are not willing to sign consent
* Children or their parents are unable to follow directions regarding gum chewing,
* Children who have a GI dysmotility disorder (e.g. chronic intestinal pseudo-obstruction)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome: first flatus, first bowel movement, first solid oral intake (any) | From time of leaving the operating room (time zero) until the time of event (first bowel movement, first flatus, first oral intake) or date of death of any cause, whichever comes first, assessed up to 30 days, measured in hours
  Documented by nurse, patient or caregiver

SECONDARY OUTCOMES:
Length of stay | From day of entering the operating room (time zero) until the time of event (day of discharge) or date of death of any cause, whichever comes first, assessed up to 30 days, measured in days
  From day admission to day of discharge
Readmission | From day of discharge (time zero) until the time of event (day of readmission) or date of death of any cause, whichever comes first, assessed up to 30 days, measured in days
  Need for readmission within 30 days of discharge
Swallowing/aspiration of gum | From day of entering the operating room (time zero) until the time of event (swallowing/aspiration of gum) or date of death of any cause, whichever comes first, assessed up to 30 days, measured as yes/no
  Measured as yes/no
Allergic reaction/adverse reaction to gum | From day of entering the operating room (time zero) until the time of event (allergic reaction/adverse reaction to gum) or date of death of any cause, whichever comes first, assessed up to 30 days, measured as yes/no
  Measured as yes/no
Re-operation | From day of entering the operating room (time zero) until the time of event (Re-operation) or date of death of any cause, whichever comes first, assessed up to 30 days, measured as yes/no
  Measured as yes/no
Need for prokinetic/anti-reflux medication | From time of leaving the operating room (time zero) until the time of event (ordering of prokinetic/anti-reflux medication) or date of death of any cause, whichever comes first, assessed up to 30days, measured in hours
  Measured as yes/no if need for additional medications to facilitate return of bowel function
Narcotic use | From time of leaving the operating room (time zero) until the time of event (ordering of narcotic medication) or date of death of any cause, whichever comes first, assessed up to 30days, measured in hours
  Quantity of narcotics consumed (mg/kg total)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Shawyer, MD, MSc, Principal Investigator — University of Manitoba
Locations (1):
- Children's Hospital of Winnipeg/Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cavusoglu YH, Azili MN, Karaman A, Aslan MK, Karaman I, Erdogan D, Tutun O. Does gum chewing reduce postoperative ileus after intestinal resection in children? A prospective randomized controlled trial. Eur J Pediatr Surg. 2009 Jun;19(3):171-3. doi: 10.1055/s-0029-1202776. Epub 2009 Apr 9. PMID 19360548
- [Result] Zhang Q, Zhao P. Influence of gum chewing on return of gastrointestinal function after gastric abdominal surgery in children. Eur J Pediatr Surg. 2008 Feb;18(1):44-6. doi: 10.1055/s-2007-989273. PMID 18302069
- [Result] Kehlet H. Fast-track surgery-an update on physiological care principles to enhance recovery. Langenbecks Arch Surg. 2011 Jun;396(5):585-90. doi: 10.1007/s00423-011-0790-y. Epub 2011 Apr 6. PMID 21468643
- [Result] Cyr C; Canadian Paediatric Society, Injury Prevention Committee. Preventing choking and suffocation in children. Paediatr Child Health. 2012 Feb;17(2):91-4. doi: 10.1093/pch/17.2.91. PMID 23372401